CLINICAL TRIAL: NCT03660098
Title: Mirror Box Therapy As a Treatment Option for Functional Movement Disorders
Acronym: MIMIC
Status: Completed | Type: Observational
Sponsor: The Cleveland Clinic (Other)
Responsible Party: Principal Investigator, Xin Xin Yu, MD, Attending Physician, The Cleveland Clinic
Other Study IDs: 18-458
Record Dates: First submitted 2018-08-08; First posted 2018-09-06 (Actual); Last update posted 2025-02-13 (Actual); Status verified 2025-02

CONDITIONS: Functional Movement Disorder
Keywords: FMD; functional movement disorder; functional neurological disorder; functional tremor; psychogenic tremor
MeSH Terms: conditions — Conversion Disorder

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

SUMMARY:
The purpose of this study is to investigate the potential of using mirror box therapy as a therapeutic technique amongst patients with functional movement disorders. It is hypothesized that a brief, single, in-office mirror therapy session will lead to a noticeable decrease in FMD-related involuntary movements.

DETAILED DESCRIPTION:
Patients diagnosed with Functional Movement Disorder presenting with a unilateral or asymmetrical bilateral hand tremor will be asked to participate in a series of hand exercises with and without a mirror box. The severity of the tremor will be rated subjectively by the subject and objectively by the neurologist after hand exercises with and without the mirror box.

ELIGIBILITY:
Inclusion Criteria:

1. Patients diagnosed with functional movement disorder by a fellowship trained movement disorders neurologist, presenting predominantly with unilateral or asymmetrical bilateral involuntary movement in the upper extremity
2. In patients with bilateral involuntary movements, the symptoms in one arm must be minimal

Exclusion Criteria:

1. Patients with moderate to severe involuntary movement in both arms
2. Significant cognitive impairment that prevents proper informed consent
3. Severe involuntary movement that interferes with the use of the apparatus
4. Patients with hemiparesis or the loss of one arm due to various reasons (e.g. amputations, birth defects, etc.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients diagnosed with functional movement disorder (functional tremor) by a fellowship trained movement disorders neurologist
Sampling Method: Probability Sample
Enrollment: 14 (Actual)
Dates: Start 2018-06-28 (Actual); Primary Completion 2022-05-17 (Actual); Study Completion 2022-05-17 (Actual)

PRIMARY OUTCOMES:
Change in Simplified Functional Movement Disorders Rating Scale (s-FMDRS) score post exercise | Because this is a one-time visit study, outcome will be measured during the visit, data reported at study conclusion after successfully recruiting 14 subjects and completing analysis with projected finish date in 1 year
  The difference in scored movement severity in the more affected hand based on the modified s-FMDRS scale during the Unified Parkinson's Disease Rating Scale (UPDRS) exam after the exercises with vs. without the mirror box. Movements are scored by video raters on a scale of 0-3, and higher score indicates more severe movement.

SECONDARY OUTCOMES:
Change in Simplified Functional Movement Disorders Rating Scale (s-FMDRS) score during exercise | Because this is a one-time visit study, outcome will be measured during the visit, data reported at study conclusion after successfully recruiting 14 subjects and completing analysis with projected finish date in 1 year
  The difference in scored movement severity in the more affected hand based on the modified s-FMDRS scale with vs. without the mirror box during exercise. Movements are scored by video raters on a scale of 0-3, and a higher score indicates more severe movement.
Change in self-perception | Because this is a one-time visit study, outcome will be measured during the visit, data reported at study conclusion after successfully recruiting 14 subjects and completing analysis with projected finish date in 1 year
  The difference in patient self-perception of movement severity based on a self-perception scale after the task with vs. without the mirror box. Patient scores movement on a scale of 0-4, with a higher score indicating more severe movement.

CONTACTS AND LOCATIONS:
Overall Officials: Xin Xin Yu, MD, Principal Investigator — The Cleveland Clinic
Locations (1):
- Cleveland Clinic, Cleveland, Ohio, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Ricciardi L, Edwards MJ. Treatment of functional (psychogenic) movement disorders. Neurotherapeutics. 2014 Jan;11(1):201-7. doi: 10.1007/s13311-013-0246-x. PMID 24356785
- [Background] Morgante F, Edwards MJ, Espay AJ. Psychogenic movement disorders. Continuum (Minneap Minn). 2013 Oct;19(5 Movement Disorders):1383-96. doi: 10.1212/01.CON.0000436160.41071.79. PMID 24092294
- [Background] Jacob AE, Kaelin DL, Roach AR, Ziegler CH, LaFaver K. Motor Retraining (MoRe) for Functional Movement Disorders: Outcomes From a 1-Week Multidisciplinary Rehabilitation Program. PM R. 2018 Nov;10(11):1164-1172. doi: 10.1016/j.pmrj.2018.05.011. Epub 2018 May 18. PMID 29783067
- [Background] Arya KN, Pandian S. Effect of task-based mirror therapy on motor recovery of the upper extremity in chronic stroke patients: a pilot study. Top Stroke Rehabil. 2013 May-Jun;20(3):210-7. doi: 10.1310/tsr2003-210. PMID 23841968
- [Background] Chan BL, Witt R, Charrow AP, Magee A, Howard R, Pasquina PF, Heilman KM, Tsao JW. Mirror therapy for phantom limb pain. N Engl J Med. 2007 Nov 22;357(21):2206-7. doi: 10.1056/NEJMc071927. No abstract available. PMID 18032777
- [Background] Moseley LG, Gallace A, Spence C. Is mirror therapy all it is cracked up to be? Current evidence and future directions. Pain. 2008 Aug 15;138(1):7-10. doi: 10.1016/j.pain.2008.06.026. Epub 2008 Jul 14. No abstract available. PMID 18621484
- [Background] Diers M, Christmann C, Koeppe C, Ruf M, Flor H. Mirrored, imagined and executed movements differentially activate sensorimotor cortex in amputees with and without phantom limb pain. Pain. 2010 May;149(2):296-304. doi: 10.1016/j.pain.2010.02.020. Epub 2010 Mar 31. PMID 20359825
- [Background] Jose N. Mirror Box Therapy. Int. J. Adv. Nur. Management. 2014 Apr;2(2):97-9.
- [Background] Chatterjee P, Banerjee R, Choudhury S, Mondal B, Kulsum MU, Chatterjee K, Kumar H. Mirror movements in Parkinson's disease: An under-appreciated clinical sign. J Neurol Sci. 2016 Jul 15;366:171-176. doi: 10.1016/j.jns.2016.05.026. Epub 2016 May 14. PMID 27288800